CLINICAL TRIAL: NCT00003528
Title: A Phase I Trial of Tomudex in Children With Leukemia
Brief Title: Raltitrexed in Treating Children With Refractory Acute Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01839; 9779; U01CA097452 (NIH); CDR0000066575 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-03-01 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — raltitrexed

ARMS (1):
- Arm I (Experimental): Patients receive raltitrexed intravenously over 15 minutes once weekly for 3 weeks followed by 1 week of rest. Treatment continues in the absence of disease progression and unacceptable toxicity.
  Interventions: Drug: raltitrexed

INTERVENTIONS:
Drug: raltitrexed — Given IV
  Other Names: D1694; ICI-D1694; TDX; Tomudex

SUMMARY:
Phase I trial to study the effectiveness of raltitrexed in treating children with refractory acute leukemia. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose and dose limiting toxicity of raltitrexed given for three weeks to children with refractory acute leukemia.

II. Determine the incidence and severity of other toxic effects of this regimen in these patients.

III. Determine a safe and tolerable dose of raltitrexed, administered in this manner, to be used in phase II studies.

IV. Determine the pharmacokinetics of this regimen in these patients. V. Determine if plasma 2' deoxyuridine concentrations are associated with raltitrexed toxicity or pharmacokinetics.

VI. Evaluate the antitumor activity of raltitrexed against recurrent leukemia.

OUTLINE: This is a dose escalation study.

Patients receive raltitrexed intravenously over 15 minutes once weekly for 3 weeks followed by 1 week of rest. Treatment continues in the absence of disease progression and unacceptable toxicity.

In the absence of dose-limiting toxicity (DLT) in the first cohort of 6 patients treated, subsequent cohorts of 6 patients each receive escalating doses of raltitrexed on the same schedule. If DLT occurs in 2 of 6 patients at a given dose level, then dose escalation ceases and the next lower dose is declared the maximum tolerated dose.

Patients are followed every 6 months for 4 years, then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven acute leukemia (M3 marrow) that is refractory to conventional therapy or for which no effective therapy exists
* No CNS leukemia
* No solid tumors
* Performance status: Karnofsky 50-100% OR Lansky at least 50 (for infants)
* Life expectancy: At least 8 weeks
* Bilirubin less than 1.5 mg/dL
* SGPT less than 5 times normal
* Normal creatinine for age OR GFR at least 70 mL/min
* No significant systemic illness such as infection
* No significant third space fluid collection
* Not pregnant or nursing
* Recovered from acute toxic effects of prior immunotherapy
* At least 6 months since prior bone marrow transplant with no evidence of graft-versus-host disease
* At least 10 days since prior biologic therapy
* At least 1 week since prior growth factors
* At least 2 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosourea) and recovered
* No concurrent steroids
* Recovered from acute toxic effects of all prior radiotherapy
* At least 2 weeks since prior local palliative radiotherapy (small port)
* At least 6 months since prior substantial bone marrow radiation
* No other concurrent anticancer therapy or investigational agents
* No concurrent nonsteroidal anti-inflammatory agents

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 1998-09; Primary Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
MTD based on incidence of DLT graded according to CTC version 2.0 | Up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven D. Weitman, Principal Investigator — Swiss Pediatric Oncology Group - Geneva
Locations (1):
- Swiss Pediatric Oncology Group - Geneva, Geneva, Switzerland